CLINICAL TRIAL: NCT00296361
Title: A Multicentre, Randomised, Open Clinical Study to Compare the Efficacy and Safety of a Combination Therapy of Tacrolimus With Sirolimus Versus Tacrolimus With Mycophenolate Mofetil in Kidney Transplantation.
Brief Title: To Compare the Efficacy and Safety of a Therapy of Tacrolimus With Sirolimus or MMF in Kidney Transplantation.
Acronym: RESTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FG-506-02-40
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Kidney Transplantation
Keywords: Tacrolimus; Kidney Transplantation; Immunosuppression; Adult; Treatment Outcomes
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Tacrolimus
- 2 (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — immunosuppression
  Other Names: Prograf, FK506

SUMMARY:
Primary objective of this study is to compare the two therapy regimens with regard to renal function by using calculated creatinine clearance. The secondary objectives are to compare the efficacy and safety profiles of the two therapy regimens.

DETAILED DESCRIPTION:
This phase III study shall provide detailed efficacy and safety information to compare this combination of sirolimus and tacrolimus with the current standard tacrolimus combination regimen (tacrolimus/MMF/steroids) which is widely used in European centres.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years of age and having end stage kidney disease who will undergo primary renal transplantation or retransplantation are eligible for the study. Patients receiving a kidney transplant, from a cadaveric or living donor (not HLA identical) with compatible AB0 blood type can be included.

Exclusion Criteria:

* Patient has a high immunological risk
* Cold ischemia time greater than 30 hours
* Patient has significant liver disease
* Patient has severe hypercholesterolaemia
* Patient is allergic or intolerant to study medication
* Patient requires ongoing dosing with corticosteroids.
* Patient or donor is known to be HIV positive
* Patient with malignancy or history of malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 634 (Actual)
Dates: Start 2004-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Renal function as assessed by calculated creatinine clearance at month 6. | 6 months

SECONDARY OUTCOMES:
Acute rejection: Incidence of and time to first acute rejection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Physician, Study Director — Astellas Pharma Europe B.V.
Locations (51):
- Australia (2):
  - Nedlands
  - Perth
- Austria (2):
  - Linz
  - Vienna
- Belgium (2):
  - Brussels
  - Leuven
- Czechia (2):
  - Olomouc
  - Ostrava
- France (6):
  - Amiens
  - Brest
  - Dijon
  - Limoges
  - Paris
  - Toulouse
- Germany (11):
  - Aachen
  - Bochum
  - Cologne
  - Freiburg im Breisgau
  - Halle
  - Hamburg
  - Hannoversch Münden
  - Hanover
  - Münster
  - Regensburg
  - Rostock
- Debrecen, Hungary
- Italy (2):
  - Milan
  - Napoli
- Rotterdam, Netherlands
- Poland (6):
  - Gdansk
  - Krakow
  - Poznan
  - Szczecin
  - Warsaw
  - Wroclaw
- Bucharest, Romania
- Spain (12):
  - Alicante
  - Badalona-Barcelona
  - Barcelona
  - Cadiz
  - Córdoba
  - Madrid
  - Málaga
  - Palma de Mallorca
  - Santander
  - Santiago de Compostela
  - Valencia
  - Valladolid
- Gothenburg, Sweden
- United Kingdom (2):
  - London
  - Nottingham

REFERENCES:
- See also: Link to FDA Website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda